CLINICAL TRIAL: NCT02112435
Title: Comparative Study of Efficacy of Titratable Mandibular Advancement Splint Versus Active Mandibular Advancement Splint to Treat Patients With Obstructive Sleep Apnea
Brief Title: Comparative Efficacy Study of Titratable Versus Active Mandibular Advancement Splint in Sleep Apnea
Acronym: SOMNYX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); University Hospital, Montpellier (Other)
Responsible Party: Principal Investigator, Nelly Huynh, Assistant research professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-011-CERES-D; NH-14SRP-Somnyx (Other: Faculté de medecine dentaire, Université de Montreal)
Record Dates: First submitted 2014-04-05; First posted 2014-04-14 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; mandibular advancement splint; active mandibular advancement splint; oral appliance
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narval ORM ® or SomnoDent ® (Active Comparator): Mandibular advancement splint (Narval ORM ® or SomnoDent ®)
  Interventions: Device: Narval ORM ® or SomnoDent ®
- Somnyx ® (Experimental): Active mandibular advancement splint (Somnyx ®)
  Interventions: Device: Somnyx ®

INTERVENTIONS:
Device: Somnyx ® — Active mandibular advancement splint
  Other Names: Active mandibular advancement appliance; Oral appliance
  Arms: Somnyx ®
Device: Narval ORM ® or SomnoDent ® — Mandibular advancement splint
  Other Names: Mandibular advancement splint; Mandibular advancement appliance; Oral appliance; Mandibular repositioning appliance; Mandibular repositioning splint
  Arms: Narval ORM ® or SomnoDent ®

SUMMARY:
Sleep apnea is a common disorder that occurs in 3-10 % of the adult population. This disorder disrupts the architecture and quality of sleep. Continuous positive airway pressure (CPAP) therapy is the standard treatment, but in some cases, it can not be used (patient refusal or intolerance). In these cases, treatment with mandibular advancement devices can bring an improvement in symptoms. Therefore, this study aims to compare the effectiveness of titratable versus active mandibular advancement splints in standard care environment. This will be based on the global response, which includes the apnea-hypopnea index and compliance in severe apnea patients who refused or where intolerant to CPAP. Following their severe apnea diagnosis and the assessment on the feasibility of placing a mandibular advancement device, follow-up visits will be scheduled after 3 months of treatment involving clinical monitoring by a physician and a dentist.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* severe OSA confirmed by polysomnography (PSG) is: 30> AHI> 15 with severe daytime sleepiness - Epworth ≥ 10 or AHI> 30
* patient in failure or refusal of CPAP treatment
* agree to participate and sign the consent form research
* speak and understand French without external assistance
* be in good health (no neurological or psychiatric syndrome).
* have a valid Social Security card (in France and Portugal only)

Exclusion Criteria:

* contra-indicated dental/periodontal states for mandibular advancement splints, such as: 1) significant edentulism (less than 3 healthy teeth / quadrant), 2) generalized periodontitis or severe parodonthopathies, 3) severe disorders of the temporomandibular joint (TMJ), 4) less than 5 mm of maximal mandibular protrusion
* dental restorations in progress or planned in the next 6 months
* psychiatric and neuromuscular disorders
* untreated cardiovascular diseases and history of stroke or myocardial infarction
* severe or morbid obesity (body mass index> 35)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Overall response rate | following 3 months of treatment
  Overall response rate (ORR) = rate of complete response (TRc) + partial response rate (PRR) =% of patients with AHI <15 or ≥ 50% reduction in AHI and compliance ≥ 5 nights / week and 5 hours / night

SECONDARY OUTCOMES:
Rate of Complete Response | following 3 months of treatment
  Rate of Complete Response (TRc) =% Patients with AHI <15 and AHI ≥ 50% reduction and compliance ≥ 5 nights / week and 5 hours / night)
Partial response rate | Following 3 months of treatment
  Partial response rate =% of patients with reduction AHI ≥ 50% with AHI> 15 or AHI <15 with reduction <50% and adherence ≥ 5 nights / week and 5 hours / night) at 3 months of treatment.
Subjective compliance | Following 3 months of treatment
  Subjective compliance
Sleep quality | Following 3 months of treatment
  sleep efficiency, total sleep time
Desaturation | Following 3 months of treatment
  desaturation index, time spent below 90%
Subjective sleep | Following 3 months of treatment
  Pittsburgh questionnaire
Quality of life | Following 3 months of treatment
  Functional outcomes sleep questionnaire (FOSQ)
Fatigue | Following 3 months of treatment
  Chalder fatigue questionnaire
Subjective daytime sleepiness | Following 3 months of treatment
  Epworth sleepiness score
Side effects | Following 3 months of treatment
  side effects and interactions with the dental evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Huynh, PhD, Principal Investigator — Université de Montréal
Locations (3):
- Université de Montréal, Montreal, Quebec, Canada
- France (2):
  - Université Montpellier, Montpellier
  - Groupe Hospitalier Pitie-Salpetriere, Paris